CLINICAL TRIAL: NCT03164577
Title: Utilizing Traditional Practices to Decrease Substance Use Among Native Americans
Brief Title: Utilizing Traditional Practices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: RAND (Other)
Responsible Party: Principal Investigator, Daniel Dickerson, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R34AA024818-01 (NIH)
Record Dates: First submitted 2017-03-27; First posted 2017-05-23 (Actual); Last update posted 2019-10-03 (Actual); Status verified 2019-10

CONDITIONS: Substance Use
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DARTNA (Active Comparator): DARTNA is a culturally-adaptable therapeutic drum behavior therapy that incorporates drumming, talking circles, and uses the 12 Steps of Alcoholics Anonymous (AA)/Narcotics Anonymous (NA) program within the conceptual framework of the Northern Plains Medicine Wheel. The Northern Plains Medicine Wheel is widely utilized as a conceptual framework and integrative approach to health and wellness for AI/ANs. This intervention consists of 12 sessions provided 2 times weekly over 6 weeks.
  Interventions: Behavioral: Drum-Assisted Recovery Therapy for Native Americans (DARTNA)
- Usual care plus (Placebo Comparator): Participants randomized to usual care plus will participate in activities for approximately the same amount of time as DARTNA participants. They will engage in health and wellness education session once weekly for 6 weeks. They will also receive care for their alcohol and other drug use, This typically consists individual counseling, group therapy, and AI/AN traditional activities in their community.
  Interventions: Other: Usual Care Plus

INTERVENTIONS:
Behavioral: Drum-Assisted Recovery Therapy for Native Americans (DARTNA) — An intervention that utilizes AI/AN drumming as its core component of treatment.
  Arms: DARTNA
Other: Usual Care Plus — Participants randomized to usual care plus will participate in activities for approximately the same amount of time as DARTNA participants. They will engage in health and wellness education session once weekly for 6 weeks. They will also receive care for their alcohol and other drug use, This typically consists individual counseling, group therapy, and AI/AN traditional activities in their community.
  Arms: Usual care plus

SUMMARY:
This study is focused on conducting a stage 1b feasibility pilot trial among 60 AI/AN men and women (for a final sample of 48 at follow-up) in an urban outpatient treatment setting to analyze the potential benefits of Drum-Assisted Recovery Therapy for Native Americans (DARTNA). Dr. Dickerson, Principal Investigator, is collaborating with Dr. Elizabeth D'Amico, co-Investigator, with Sacred Path Indigenous Wellness Center, a community-based organization providing consultative services for American Indians/Alaska Natives (AI/ANs).

A feasibility randomized clinical trial will be conducted within an urban setting and will compare urban AI/AN males and females with AOD disorders who receive DARTNA (n=30) to AI/AN males and females with AOD disorders who receive usual care plus (n=30). Compare outcomes at end of treatment and 3-months post-treatment to gather data that can be used to judge the feasibility of a larger trial, and to plan that trial. Obtain information on (a) clinically significant changes in AOD use, (b) clinically significant changes in mental health, physical health, spirituality, cognition, adoption of 12-step principles and practices, and cultural identification, and (c) estimate covariate correlations, reliability of measures and likely effect sizes.

DETAILED DESCRIPTION:
Alcohol and other drug (AOD) abuse among American Indians and Alaska Natives (AI/ANs) is a significant health issue in the United States as rates of AOD use among AI/ANs have continually been high since national data were collected among AI/ANs beginning in the 1980's. In 2013, AI/ANs had the highest rate of AOD dependence and abuse compared with other racial groups.

However, very few AOD abuse treatments utilizing traditional based healing, such as drumming, have undergone rigorous scientific research. Drum-Assisted Recovery Therapy for Native Americans (DARTNA) is a new AOD use intervention integrating AI/AN drumming, 12-step philosophy, and concepts focused on the Medicine Wheel. In a recently completed National Center for Complementary and Alternative Medicine (NCCAM)-funded study (R21AT005360), the PI completed key components of DARTNA development (stage 1a) including demonstrating feasibility and acceptability, establishing procedures for therapist adherence procedures, developing a treatment manual, and conducting a pretest among ten AI/AN men (n=5) and women (n=5) with promising preliminary findings.

This study is focused on conducting a stage 1b feasibility pilot trial among 60 AI/AN men and women (for a final sample of 48 at follow-up) in an urban outpatient treatment setting to analyze the potential benefits of Drum-Assisted Recovery Therapy for Native Americans (DARTNA). Dr. Dickerson, Principal Investigator, is collaborating with Dr. Elizabeth D'Amico, co-Investigator, with Sacred Path Indigenous Wellness Center, a community-based organization providing consultative services for American Indians/Alaska Natives (AI/ANs).

ELIGIBILITY:
Inclusion Criteria:

1) self-identify as AI/AN male or female, (2) be seeking treatment for their drug or alcohol dependence; (3) be 18-59 years of age or older; (4) meet Diagnostic and Statistical Manual of Mental Disorders-Fourth Edition (Text Revision) (DSM-IV-TR) criteria for AOD use disorders;

Exclusion Criteria:

1. have a mental health or medical history that, in the judgment of the study physician or PI, show no clinically significant contraindications for study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — 30 males and 30 females
Enrollment: 62 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-02-20 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Change in alcohol and other drug use based on the Timeline Follow Back | Change from baseline alcohol and other drug use at end of treatment (42-72 days) and at 3-month follow-up (132-177 days)
  recent alcohol and other drug use will be tracked

SECONDARY OUTCOMES:
Change in physical health status utilizing the Physical health questionnaire (PHQ) | Change from baseline physical health status at end of treatment (42-72 days) and at 3-month follow-up (132-177 days)
  This assessment is a brief self-report scale of somatic symptoms.
Change in Spirituality utilizing the Functional Assessment of Chronic Illness Therapy (FACIT): Spiritual Questions Only-Expanded | Change from baseline spirituality at end of treatment (42-72 days) and at 3-month follow-up (132-177 days)
  This 23-item spirituality scale measures comfort and strength derived from one's spiritual beliefs or connection to God or a Higher Power.
Change in cognitive function utilizing the Functional Assessment of Cancer Therapy-Cognitive Function (FACT-Cog), Version 3 | Change from baseline cognitive function at end of treatment (42-72 days) and at 3-month follow-up (132-177 days)
  This 37-item cognitive function scale measures areas associated with cognitive function, including perceived cognitive impairments, comments from others (i.e., observations by others regarding cognition), perceived cognitive abilities, and impact on quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- United American Indian Involvement, Inc., Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No